CLINICAL TRIAL: NCT02313272
Title: A Phase I Trial of Hypofractionated Stereotactic Irradiation (HFSRT) With Pembrolizumab and Bevacizumab in Patients With Recurrent High Grade Gliomas
Brief Title: Hypofractionated Stereotactic Irradiation (HFSRT) With Pembrolizumab and Bevacizumab for Recurrent High Grade Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17978
Record Dates: First submitted 2014-12-05; First posted 2014-12-10 (Estimated); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-12

CONDITIONS: Malignant Glioma
Keywords: neoplasms; high-grade glioma; recurrent glioma; glioma; Hypofractionated Stereotactic Irradiation (HFSRT); Bevacizumab; Pembrolizumab; recurrent high-grade glioma; Grade III malignant glioma; Grade IV malignant glioma; brain and nervous system
MeSH Terms: conditions — Glioma; Neoplasms; Neurologic Manifestations | interventions — pembrolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HFSRT with Pembrolizumab and Bevacizumab (Experimental): Hypofractionated Stereotactic Irradiation (HFSRT). Pembrolizumab intravenous (IV) infusion every 3 weeks. Bevacizumab administered intravenously every 2 weeks.
  Interventions: Radiation: Hypofractionated Stereotactic Irradiation (HFSRT); Drug: Pembrolizumab; Drug: Bevacizumab

INTERVENTIONS:
Radiation: Hypofractionated Stereotactic Irradiation (HFSRT) — Radiation therapy treatment (FSRT) which will be given to participants over 5 days.
Drug: Pembrolizumab — Dose Escalation: The dose of pembrolizumab will be escalated per schema in a 3+3 fashion. The starting dose (i.e., dose level 1) will be 100 mg.
  Dose Expansion: The pembrolizumab dose used in the dose expansion cohort will be maximum tolerated dose (MTD) determined from the dose escalation phase.
  Other Names: Keytruda®; MK-3475
Drug: Bevacizumab — Initial cycle of bevacizumab must start within 10 days of registering to the trial. It will be given concurrent with radiation therapy. Bevacizumab will be administered intravenously at a dose of 10 mg/kg every 2 weeks. Doses will be adjusted if there is a > 10% change in weight.
  Other Names: Avastin®

SUMMARY:
The purpose of this study is to see if the addition of the investigation drug called pembrolizumab (Keytruda®) to radiation therapy and bevacizumab (Avastin®) is safe and can help with controlling the growth of tumors, in participants with recurrent high grade glioma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of World Health Organization (WHO) Grade III (except anaplastic oligodendroglioma) or IV malignant glioma.
* Documented recurrence by diagnostic biopsy or contrast enhanced magnetic resonance imaging (MRI) performed within 28 days of entry into the trial as per Response Assessment Criteria for High-Grade Gliomas (RANO) Criteria.
* Patients with recurrent WHO Grade III gliomas should have received one prior treatment for recurrent high grade disease.
* Maximum diameter of enhancing tumor (target lesion) should be ≤ 3.5 cm.
* Interval of ≥ 6 months after the end of prior radiation therapy is required unless there is a new recurrence outside of the previous radiotherapy treatment field.
* Previous first line treatment with at least standard dose of radiotherapy (total dose ≥ 54 Gy) and temozolomide.
* Interval of ≥ 4 weeks since surgical resection prior to entry into the trial.
* Interval of ≥ 4 weeks after last administration of any investigational agent or prior cytotoxic therapy (except bevacizumab). There should be 14 days interval between the last dose of bevacizumab and first day of treatment on study.
* Age 18 years or older on day of signing informed consent.
* Karnofsky performance status ≥ 70.
* Demonstrate adequate organ function.
* Resting baseline O2 saturation by pulse oximetry of ≥ 92% at rest.
* Must have recovered from the toxic effects of prior therapies.
* Willing and able to provide written informed consent/assent for the trial.
* Life expectancy ≥ 12 weeks.
* Female participants of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving first dose of study medication. Must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.
* Male participants should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* More than 3 recurrences of high grade glioma.
* Has anaplastic oligodendroglioma.
* Has received reradiation to recurrent disease (other than standard frontline adjuvant radiation therapy).
* Recurrent tumors near the brainstem and optic chiasm must not have received prior radiation therapy.
* Infratentorial, or leptomeningeal evidence of recurrent disease.
* Recurrent or persistent tumor (enhancing area) greater than 3.5 cm in maximum diameter.
* Prior treatment with Gliadel unless it was administered as first line treatment and ≥ 3 months prior to study treatment.
* Unable (due to existent medical condition) or unwilling to have a contrast enhanced MRI of brain.
* Currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of first dose of treatment.
* Diagnosis of immunodeficiency or is receiving systemic immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Physiologic doses of steroid therapy (≤ 10 mg/day prednisone equivalents) is allowed.
* Prior chemotherapy, targeted small molecule therapy, or monoclonal antibody (except bevacizumab) within 4 weeks prior to study Day 1 or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier. Wash out period for bevacizumab is 14 days.
* Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Active autoimmune disease requiring systemic treatment within past 3 months or documented history of clinically severe autoimmune disease, or syndrome that requires systemic steroids or immunosuppressive agents.
* Evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Active infection requiring systemic therapy.
* Prior allergic reaction to Bevacizumab.
* History of uncontrolled hypertension, hypertensive crisis or hypertensive encephalopathy.
* History of a non-healing wound, ulcer, or bone fracture within 90 days (3 months) prior to entry into the trial.
* History of gastrointestinal bleeding or any other hemorrhage/bleeding event ≥ grade 3 (CTCAE, v. 4) within 30 days prior to entry in to the trial.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 1 of treatment on study.
* Requires escalating or chronic supraphysiologic doses of corticosteroids (> 10 mg/day prednisone equivalents).
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Prior therapy with an anti-Programmed Death 1(PD-1), anti-Programmed Death-1 Ligand 1 (PD-L1), anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Known active Hepatitis B.
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2021-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Solmaz Sahebjam, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Bruningk SC, Peacock J, Whelan CJ, Brady-Nicholls R, Yu HM, Sahebjam S, Enderling H. Intermittent radiotherapy as alternative treatment for recurrent high grade glioma: a modeling study based on longitudinal tumor measurements. Sci Rep. 2021 Oct 12;11(1):20219. doi: 10.1038/s41598-021-99507-2. PMID 34642366

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: HFSRT With Pembrolizumab and Bevacizumab: Hypofractionated Stereotactic Irradiation (HFSRT) radiation therapy treatment (FSRT) given to participants over 5 days. 100 mg Pembrolizumab intravenous (IV) infusion every 3 weeks. 10 mg/kg Bevacizumab administered intravenously every 2 weeks.
- Dose Level 2: HRSRT With Pembrolizumb and Bevacizumab; Participants Treated at Maximum Tolerated Dose: Hypofractionated Stereotactic Irradiation (HFSRT) radiation therapy treatment (FSRT) given to participants over 5 days. 200 mg Pembrolizumab intravenous (IV) infusion every 3 weeks. 10 mg/kg Bevacizumab administered intravenously every 2 weeks.
Period: Overall Study
Arm/Group | Dose Level 1: HFSRT With Pembrolizumab and Bevacizumab | Dose Level 2: HRSRT With Pembrolizumb and Bevacizumab | Participants Treated at Maximum Tolerated Dose
Started | 3 | 16 | 13
Completed | 3 | 16 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: HFSRT With Pembrolizumab and Bevacizumab | Dose Level 2: HRSRT With Pembrolizumb and Bevacizumab | Participants Treated at Maximum Tolerated Dose | Total
Number analyzed (Participants) | 3 | 16 | 13 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 14 | 11 | 28
  >=65 years | 0 | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 5 | 11
  Male | 3 | 10 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 2 | 15 | 12 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 15 | 13 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 16 | 13 | 32

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The pembrolizumab dose used in the dose expansion cohort will be MTD determined from the dose escalation phase. Dose Escalation: The maximum tolerated dose (MTD) is the highest dose of pembrolizumab in combination with bevacizumab after radiation therapy that does not cause unacceptable toxicity in more than one of six patients at that dose level. The MTD is defined as one dose level below the highest toxic dose (i.e., the Dose Limiting Toxicity (DLT) dose).
Time Frame: Up to 24 months
Population: Participants in dose finding phase of study
Measure: Number; unit: mg
Groups:
- HFSRT With Pembrolizumab and Bevacizumab: Hypofractionated Stereotactic Irradiation (HFSRT). Pembrolizumab intravenous (IV) infusion every 3 weeks. Bevacizumab administered intravenously every 2 weeks.
  Hypofractionated Stereotactic Irradiation (HFSRT): Radiation therapy treatment (FSRT) which will be given to participants over 5 days.
  Pembrolizumab: Dose Escalation: The dose of pembrolizumab will be escalated per schema in a 3+3 fashion. The starting dose (i.e., dose level 1) will be 100 mg.
  Dose Expansion: The pembrolizumab dose used in the dose expansion cohort will be maximum tolerated dose (MTD) determined from the dose escalation phase.
  Bevacizumab: Initial cycle of bevacizumab must start within 10 days of registering to the trial. It will be given concurrent with radiation therapy. Bevacizumab will be administered intravenously at a dose of 10 mg/kg every 2 weeks. Doses will be adjusted if there is a > 10% change in weight.
Arm/Group | HFSRT With Pembrolizumab and Bevacizumab
Number analyzed (Participants) | 19
mg | 200

2. Secondary Outcome: Response Rate (RR)
Description: Response rate of pembrolizumab given in combination with bevacizumab and hypofractionated stereotactic re-irradiation of recurrent high grade gliomas. Response to treatment will be assessed by the investigator and according to the Response Assessment Criteria for High-Grade Gliomas (RANO Criteria). Brain MRI will be performed every 6 weeks beginning at the end of Week 6 (± 1 week) for 3 cycles and then every 12 weeks (± 1 week) until disease progression or treatment discontinuation, whichever occurs later.
Time Frame: Up to 24 months
Population: All participants who received at least one dose of study drugs
Measure: Number; unit: percentage of participants
Arm/Group | Dose Level 1: HFSRT With Pembrolizumab and Bevacizumab | Dose Level 2: HRSRT With Pembrolizumb and Bevacizumab | Participants Treated at Maximum Tolerated Dose
Number analyzed (Participants) | 3 | 16 | 13
percentage of participants
  Complete Response | 33.33 | 6.25 | 0
  Partial Response | 33.33 | 62.5 | 71.88

ADVERSE EVENTS:
Time Frame: Adverse events recorded day 1 of study treatment through 30 days following cessation of treatment, 37 months in total.
Arm/Group | Dose Level 1: HFSRT With Pembrolizumab and Bevacizumab | Dose Level 2: HRSRT With Pembrolizumb and Bevacizumab | Participants Treated at Maximum Tolerated Dose
All-Cause Mortality (participants affected / at risk) | 3/3 | 14/16 | 10/13
Serious Adverse Events (participants affected / at risk) | 3/3 | 7/16 | 8/13
Other Adverse Events (participants affected / at risk) | 3/3 | 16/16 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: HFSRT With Pembrolizumab and Bevacizumab (N=3) | Dose Level 2: HRSRT With Pembrolizumb and Bevacizumab (N=16) | Participants Treated at Maximum Tolerated Dose (N=13)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (2) | 2 (3)
Wound infection (Infections and infestations) | 0 (0) | 3 (6) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures-Other (Surgical and medical procedures) | 2 (2) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified -Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness, right sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous System disorders- Other (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Shunt placement surgery
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3)
Psychiatric disorders - Other (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Lung infection - pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders -Other (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — double vision
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Facial muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Muscle Weakness - Left Side
Nervous System disorders -Other (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalitis Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: HFSRT With Pembrolizumab and Bevacizumab (N=3) | Dose Level 2: HRSRT With Pembrolizumb and Bevacizumab (N=16) | Participants Treated at Maximum Tolerated Dose (N=13)
Hallucinations (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 4 (7) | 3 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (22) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 5 (6)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 3 (3)
Ataxia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (4) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (2) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 3 (4) | 2 (3)
Cholesterol high (Investigations) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 2 (3) | 7 (10)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 3 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (2) | 4 (5) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 5 (6) | 5 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 1 (2) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 3 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (2) | 1 (1) | 2 (4)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 6 (7) | 3 (5)
Fatigue (General disorders) | 1 (2) | 7 (9) | 5 (8)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 4 (6) | 4 (8)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 2 (4)
Gait disturbance (General disorders) | 1 (1) | 5 (5) | 4 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Excess saliva
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6) | 4 (5)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (5) | 8 (10)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 3 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 7 (12) | 7 (9)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (10) | 1 (1)
Hypertension (Vascular disorders) | 2 (4) | 3 (3) | 5 (11)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 4 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (3) | 4 (5)
Infections and infestations -Other (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Mediport infection
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (3)
IVth nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Localized edema (General disorders) | 0 (0) | 2 (4) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (3)
Lymphocyte count decreased (Investigations) | 1 (1) | 7 (21) | 9 (15)
Memory impairment (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (8) | 5 (5)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) — benign neoplasm left eye
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 3 (5) | 3 (5)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (3)
Pain (General disorders) | 0 (0) | 6 (7) | 4 (5)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2)
Platelet count decreased (Investigations) | 2 (4) | 5 (9) | 3 (5)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (2) | 6 (9) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Psychiatric disorders - Other (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) — panic attacks
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 3 (3) | 3 (5) | 3 (5)
Sinus pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (5) | 3 (4)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2) | 2 (3)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (4) | 1 (1)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 2 (21) | 1 (6)
White blood cell decreased (Investigations) | 0 (0) | 3 (4) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1) | 0 (0) | 2 (2) — Right parietal stereotactic resection of tumor
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 3 (11) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (2) | 2 (2)
Intraoperative musculoskeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other (Investigations) | 0 (0) | 0 (0) | 1 (1) — Hyperammonemia
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Nose bleeds

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT02313272/Prot_SAP_000.pdf